CLINICAL TRIAL: NCT04689386
Title: Efecto De La Fisioterapia Respiratoria Sobre El Desarrollo De Niños/as Prematuros. Estudio Longitudinal.
Brief Title: Effect of Chest Physiotherapy on the Development of Preterm Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Collaborators: Fundación para la Salud Infantil de la Comunidad Valenciana (Unknown)
Responsible Party: Principal Investigator, Ana Igual Blasco, Degree in Physiotherapy, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 74244433
Record Dates: First submitted 2020-10-02; First posted 2020-12-30 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: Development, Infant; Respiratory Distress Syndrome in Premature Infant
Keywords: Premature Infant; Respiratory Distress Syndrome; Chest Physiotherapy; Development
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I Stimulation of "reflex rolling" from the Vojta method (Experimental)
  Interventions: Other: Group I (GE-I) - Stimulation of "reflex rolling" from the Vojta method
- Group II Expiratory flow increase technique (Experimental)
  Interventions: Other: Group II (GE-II) - expiratory flow increase technique
- Control Group (No Intervention): Routine intervention in the NICU with mechanical ventilation.

INTERVENTIONS:
Other: Group I (GE-I) - Stimulation of "reflex rolling" from the Vojta method — This manoeuvre does not require the newborn to be moved, but only a slight rotation of the head towards the side from which the stimulus is delivered. The starting position for performing the first phase of reflex rolling is the asymmetric supine position, with the limbs freely lying on the resting surface.
  A digital pressure will exert on the chest area, where the mammillary line crosses the insertion of the diaphragm, either at the level of the 6th rib, or between the 5th and the 6th, or between the 6th and the 7th. A one minute stimulus will be performed on each side. The intervention will be repeated twice a day, ensuring that the period between one intervention and another is at least two hours.
  Arms: Group I Stimulation of "reflex rolling" from the Vojta method
Other: Group II (GE-II) - expiratory flow increase technique — The technique adapted to the premature infant will be performed. This maneuver consists of slowly applying light pressure to the infant's chest with one hand, obliquely, starting from the end of the inspiratory plateau until the end of expiration, which is prolonged. The hand should be placed between the sternal notch and the xiphoid process of the newborn's sternum. The therapist's other hand is placed on the last ribs (without applying pressure) as a bridge, of which the columns are the thumb and forefinger (or middle finger). Therefore, contact with the infant's abdomen is avoided and the expansion of the lower rib is limited, allowing a better displacement of the diaphragm and avoiding an increase in intra-abdominal pressure. The maneuver will be repeated three times, respecting the infant's responses and their physiological constants. The intervention will be repeated twice a day, trying to ensure that the period between one intervention and another is at least 2 hours.
  Arms: Group II Expiratory flow increase technique

SUMMARY:
The aim of this study is to investigate the effect of the stimulation of "reflex rolling" from the Vojta method and the effect of the expiratory flow increase technique on the development of the preterm infants. In the same way, it will be assessed whether the application of these techniques produce pain.

This application will be carried out in preterm infants of less than 32 weeks of gestation with neonatal respiratory distress syndrome (SDR) and carriers of mechanical ventilation. The intervention will take place in the neonatal intensive care unit (NICU) The intervention period is one month (4 weeks) and different follow-ups will be carried out at term age, at 3, 6, 9 and 12 months of corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infants <32 gestational age
* Admitted to the NICU
* With SDR
* Hemodynamically stable
* Stable convulsive pictures
* Controlled thermoregulation
* Mechanical ventilation (invasive or non-invasive)
* Parents / guardians of legal age, with sufficient cognitive ability to understand consent
* Signature of consent

Exclusion Criteria:

* Periventricular leukomalacia
* Grade III and IV intraventricular hemorrhage
* Rib fracture
* Asphyxia at birth
* Necrotizing enterocolitis > or = II B

Abandoned Criteria:

* Appearance of any of the complications mentioned above
* Hospital transfer
* Hospital discharge (if the intervention at home cannot be followed)
* Voluntary decision of parents / guardians to abandon the study
* Medical decision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of change in motor development with Bayley III scale at 3, 6, 9 and 12 months of corrected age | at 3, 6, 9 and 12 months of corrected age.
  The motor area of the Bayley III scale will be measured at 3, 6, 9 and 12 months of corrected age. The motor scale has two subscales, the gross motor scale and the fine motor scale. This motor scale is made up of 138 items (the gross motor scale is made up of 72 items and the fine motor scale of 66 items) through which it evaluates the degree of body control, coordination of large muscle masses and skill manipulative of hands and fingers.

SECONDARY OUTCOMES:
Motor activity of the premature infant measured through the Alberta Infant Motor Scale (AIMS) at term age, at 3, 6, 9 and 12 months of corrected age | at term age, at 3, 6, 9 and 12 months of corrected age.
  Alberta Infant Motor Scale consists of 58 items based on descriptions of postural control in supine decubitus (9 items), prone decubitus (21 items), sitting (12 items) and standing (16 items). It is designed for children from 0 to 18 months.
Pain during the intervention measured through the PIPP scale | Daily in all interventions, that is, every day that the intervention is applied during the month of the intervention period
  The Premature Infant Pain Profile (PIPP) scale is based on mixed behavioral and physiological indicators. It has seven items and each item will be estimated from 0 to 3 to assess pain in premature infants.
  The maximum score is 21, and in term newborns it is 18. According to the score obtained, it is concluded:
  * Minimal pain or no pain: 0 to 6 points
  * Moderate pain: 7 to 12 points
  * Intense or severe pain: if it is greater than 12 points
Measurements related to lung function (PaO2 and PaCO2 or PvO2 and PvO2) | The measurement performed by the neonatal service will be recorded. It will be recorded in the first assessment, in the final assessment (the day after finishing the intervention) and daily during the month of the intervention period
  Pa02 and PaCO2 or PvO2 and PvO2 will be assessed with an arterial blood gas / arterialized blood / venous blood gas from the measurement carried out by the neonatal service. It will be recorded in the first evaluation, in the final evaluation (the day after finishing the intervention) and daily during the intervention.
Measurements related to lung function (SatO2) | The day of the initial and final evaluation (the day after finishing the intervention) in the three groups. In addition, they will be measured before and after each intervention in GE-I and GE-II during the month that the intervention lasts.
  Sat02 and will be measured with the pulse oximeter.
Measurements related to lung function (respiratory rate) | From date of randomization until 1 month
  The values of respiratory rate will be those rebounded by mechanical ventilation or pulse oximeter.
Measurements related to lung function (FiO2) | From date of randomization until 1 month
  The values of FiO2 will be those rebounded by mechanical ventilation
Measurements related to lung function (PEEP and PIP) | From date of randomization until 1 month
  The values of PEEP and PIP will be those rebounded by mechanical ventilation
Heart rate | From date of randomization until 1 month
  Heart rate will be measured with the pulse oximeter.
Injury or respiratory failure | From date of randomization until 1 month
  Injury or respiratory failure will be calculated using the following formula: PaO2 / FiO2
Days of contribution of 02 | From date of randomization until hospital discharge. This value will not be complete until the end of the intervention in all cases, an average of around 1 year
  The days of contribution of 02 greater than 21% will be collected from the clinical history.
Days of mechanical ventilation. | From date of randomization until hospital discharge. This value will not be complete until the end of the intervention in all cases, an average of around 1 year
  The days of mechanical ventilation will be collected from the clinical history.
Start time of autonomous feeding | At hospital discharge.
  The age of the premature infant at the time of initiation of autonomous feeding will be collected from the clinical history.
Hospitalization time | At hospital discharge.
  The days of hospitalization will be collected from the clinical history.
Anthropometric measures | They will be measured at the initial assessment (the day before the start of the intervention), at the final assessment after the intervention period, and at hospital discharge.
  The weight measurement will be done through a scale or through the clinical history. Measurement of height and head circumference will be done with a tape measure or through the clinical history.
Weight | They will be measured at the initial assessment (the day before the start of the intervention), at the final assessment (after the intervention period), and at hospital discharge.
  The weight measurement will be done through a scale or through the clinical history.
Height | They will be measured at the initial assessment (the day before the start of the intervention), at the final assessment (after the intervention period), and at hospital discharge.
  Measurement of height will be done with a tape measure or through the clinical history.
cephalic perimeter | They will be measured at the initial assessment (the day before the start of the intervention), at the final assessment (after the intervention period), and at hospital discharge.
  Measurement cephalic perimeter will be done with a tape measure or through the clinical history.
Family and personal history | First day of participation in the study
  A semi-structured interview will record the history of the pregnancy (type of fertilization: natural or artificial; parity: single, twin, multiple; type of delivery: eutocic, dystocic, etc.) and family data (type of family, age of the mother / father, educational level, socioeconomic level, etc.).
  Gestational age, gender, and APGAR score will be recorded from medical clinica.
Numbers of hospital admissions for respiratory infection up to 12 months of corrected age | Assessment of 12 months of corrected age.
  The numbers of hospital admissions for respiratory infection up to 12 months of corrected age will be recorded through a questionnaire that will be delivered to the family.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Torrecárdenas, Almería, Almería
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abman SH, Bancalari E, Jobe A. The Evolution of Bronchopulmonary Dysplasia after 50 Years. Am J Respir Crit Care Med. 2017 Feb 15;195(4):421-424. doi: 10.1164/rccm.201611-2386ED. No abstract available. PMID 28199157
- [Background] Agerholm H, Rosthoj S, Ebbesen F. Developmental problems in very prematurely born children. Dan Med Bull. 2011 Jun;58(6):A4283. PMID 21651878
- [Background] Bancalari E, Jain D. Bronchopulmonary Dysplasia: 50 Years after the Original Description. Neonatology. 2019;115(4):384-391. doi: 10.1159/000497422. Epub 2019 Apr 11. PMID 30974430
- [Background] Baker CD, Abman SH. Impaired pulmonary vascular development in bronchopulmonary dysplasia. Neonatology. 2015;107(4):344-51. doi: 10.1159/000381129. Epub 2015 Jun 5. PMID 26044102
- [Background] Baker CD, Abman SH, Mourani PM. Pulmonary Hypertension in Preterm Infants with Bronchopulmonary Dysplasia. Pediatr Allergy Immunol Pulmonol. 2014 Mar 1;27(1):8-16. doi: 10.1089/ped.2013.0323. PMID 24669351
- [Background] Bayley, N. (2015). Escala Bayley de desarrollo infantil -III (Bayley-III). España: Person Educación
- [Background] Camy LF, Mezzacappa MA. Expiratory flow increase technique and acid esophageal exposure in infants born preterm with bronchopulmonary dysplasia. Pediatr Phys Ther. 2011 Winter;23(4):328-33. doi: 10.1097/PEP.0b013e31823565c3. PMID 22090070
- [Background] Cohen, J. (1988). Statistical Power Analysis for the Behavioral Sciences. 2nd. edit., Hillsdale, N.J., Erlbaum (Primera edición, 1977 New York: Academic Press)
- [Background] Davidson J, Garcia KM, Yi LC, Goulart AL, Santos AM. Prevalence and factors associated with thoracic alterations in infants born prematurely. Rev Assoc Med Bras (1992). 2012 Nov-Dec;58(6):679-84. PMID 23250096
- [Background] Fernández Rego, F. J. y Gómez-Conesa, A. (2014). Importancia del tratamiento de Fisioterapia en el síndrome de dificultad respiratoria y en la displasia broncopulmonar. Fisioterapia, 245-246. https://doi.org/10.1016/j.ft.2014.09.004
- [Background] Gasquez Góngora, JJ. (2010). Displasia broncopulmonar. Revista mexicana de Pediatría, 77(1), 27-31.
- [Background] Giannantonio C, Papacci P, Ciarniello R, Tesfagabir MG, Purcaro V, Cota F, Semeraro CM, Romagnoli C. Chest physiotherapy in preterm infants with lung diseases. Ital J Pediatr. 2010 Sep 26;36:65. doi: 10.1186/1824-7288-36-65. PMID 20868518
- [Background] Gómez Conesa, A., Fernández-Rego, F.J., y Agueras Arenas, J.J. (2016). Vojta therapy in the reduction of perinatal risk in preterm infants with respiratory distress syndrome and bronchopulmonary dysplasia. Physiotherapy, 102, 199. DOI:https://doi.org/10.1016/j.physio.2016.10.242
- [Background] Gonzáalvez Armengod, C., Omaña Alonso, MF. (2006). Protocolos de Neonatología: Síndrome de diestrés respiratorio neonatal o enfermedad de membrana hialina. Bol Pediatr, 46 (1), 160-165.
- [Background] Hestnes J, Hoel H, Risa OJ, Romstol HO, Roksund O, Frisk B, Thorsen E, Halvorsen T, Clemm HH. Ventilatory Efficiency in Children and Adolescents Born Extremely Preterm. Front Physiol. 2017 Jul 13;8:499. doi: 10.3389/fphys.2017.00499. eCollection 2017. PMID 28751866
- [Background] Islam JY, Keller RL, Aschner JL, Hartert TV, Moore PE. Understanding the Short- and Long-Term Respiratory Outcomes of Prematurity and Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2015 Jul 15;192(2):134-56. doi: 10.1164/rccm.201412-2142PP. PMID 26038806
- [Background] Lapcharoensap W, Gage SC, Kan P, Profit J, Shaw GM, Gould JB, Stevenson DK, O'Brodovich H, Lee HC. Hospital variation and risk factors for bronchopulmonary dysplasia in a population-based cohort. JAMA Pediatr. 2015 Feb;169(2):e143676. doi: 10.1001/jamapediatrics.2014.3676. Epub 2015 Feb 2. PMID 25642906
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Lean RE, Han RH, Smyser TA, Kenley JK, Shimony JS, Rogers CE, Limbrick DD Jr, Smyser CD. Altered neonatal white and gray matter microstructure is associated with neurodevelopmental impairments in very preterm infants with high-grade brain injury. Pediatr Res. 2019 Sep;86(3):365-374. doi: 10.1038/s41390-019-0461-1. Epub 2019 Jun 18. PMID 31212303
- [Background] Morales, M. S. L., Grenfell, A. M. G., Vargas, M. P. S., y Ramos, J. D. T. (2008). La nueva displasia broncopulmonar. Parte I. Revista del Instituto Nacional de Enfermedades Respiratorias, 21(3), 221-234.
- [Background] Pandya YS, Shetye J, Nanavati R, Mehta A. Resolution of lung collapse in a preterm neonate following chest physiotherapy. Indian J Pediatr. 2011 Sep;78(9):1148-50. doi: 10.1007/s12098-011-0397-x. Epub 2011 Mar 9. PMID 21390521
- [Background] Pallás, C., Cruz, J., y Medina, C. (2001). Apoyo al desarrollo de los niños nacidos demasiado pequeños, demasiado pronto. Madrid: Ministerio de trabajo y asuntos sociales. Documentos 56/2000. Real Patronato sobre discapacidad.
- [Background] Perez Tarazona S, Rueda Esteban S, Alfonso Diego J, Barrio Gomez de Aguero MI, Callejon Callejon A, Cortell Aznar I, de la Serna Blazquez O, Domingo Miro X, Garcia Garcia ML, Garcia Hernandez G, Luna Paredes C, Mesa Medina O, Moreno Galdo A, Moreno Requena L, Perez Perez G, Salcedo Posadas A, Sanchez Solis de Querol M, Torrent Vernetta A, Valdesoiro Navarrete L, Vilella Sabate M; el Grupo de Trabajo de Patologia Respiratoria Perinatal de la Sociedad Espanola de Neumologia Pediatrica. [Guidelines for the follow up of patients with bronchopulmonary dysplasia]. An Pediatr (Barc). 2016 Jan;84(1):61.e1-9. doi: 10.1016/j.anpedi.2015.04.020. Epub 2015 Jun 15. Spanish. PMID 26089228
- [Background] Piper, M. C., & Darrah, J. (1994). Motor assesssment of the developing infant. Recuperado de https://www.fylkesmannen.no/contentassets/880e78d8d11e415eb33008d556107d69/motor-assesssment-of-the-developing-infant---ellen-roseth.pdf
- [Background] Salcedo Posadas, A., González, E., Herráiz, R., y Rodriguez Cimadevilla, J.L. (2014). Normas para control y seguimiento de niños con displasia broncopulmonar (enfermedad pulmonar crónica en la infancia). Salud(i)Ciencia, 20, 730-737.
- [Background] Sanchez Luna M, Moreno Hernando J, Botet Mussons F, Fernandez Lorenzo JR, Herranz Carrillo G, Rite Gracia S, Salguero Garcia E, Echaniz Urcelay I; Comision de Estandares de la Sociedad Espanola de Neonatologia. [Bronchopulmonary dysplasia: definitions and classifications]. An Pediatr (Barc). 2013 Oct;79(4):262.e1-6. doi: 10.1016/j.anpedi.2013.02.003. Epub 2013 Apr 10. Spanish. PMID 23582451
- [Background] Simpson SJ, Logie KM, O'Dea CA, Banton GL, Murray C, Wilson AC, Pillow JJ, Hall GL. Altered lung structure and function in mid-childhood survivors of very preterm birth. Thorax. 2017 Aug;72(8):702-711. doi: 10.1136/thoraxjnl-2016-208985. Epub 2017 Jan 24. PMID 28119488
- [Background] Sonnenschein-van der Voort AM, Arends LR, de Jongste JC, Annesi-Maesano I, Arshad SH, Barros H, Basterrechea M, Bisgaard H, Chatzi L, Corpeleijn E, Correia S, Craig LC, Devereux G, Dogaru C, Dostal M, Duchen K, Eggesbo M, van der Ent CK, Fantini MP, Forastiere F, Frey U, Gehring U, Gori D, van der Gugten AC, Hanke W, Henderson AJ, Heude B, Iniguez C, Inskip HM, Keil T, Kelleher CC, Kogevinas M, Kreiner-Moller E, Kuehni CE, Kupers LK, Lancz K, Larsen PS, Lau S, Ludvigsson J, Mommers M, Nybo Andersen AM, Palkovicova L, Pike KC, Pizzi C, Polanska K, Porta D, Richiardi L, Roberts G, Schmidt A, Sram RJ, Sunyer J, Thijs C, Torrent M, Viljoen K, Wijga AH, Vrijheid M, Jaddoe VW, Duijts L. Preterm birth, infant weight gain, and childhood asthma risk: a meta-analysis of 147,000 European children. J Allergy Clin Immunol. 2014 May;133(5):1317-29. doi: 10.1016/j.jaci.2013.12.1082. Epub 2014 Feb 12. PMID 24529685
- [Background] Srinivasan L, Dutta R, Counsell SJ, Allsop JM, Boardman JP, Rutherford MA, Edwards AD. Quantification of deep gray matter in preterm infants at term-equivalent age using manual volumetry of 3-tesla magnetic resonance images. Pediatrics. 2007 Apr;119(4):759-65. doi: 10.1542/peds.2006-2508. PMID 17403847
- [Background] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730
- [Background] Stoll BJ, Hansen NI, Bell EF, Walsh MC, Carlo WA, Shankaran S, Laptook AR, Sanchez PJ, Van Meurs KP, Wyckoff M, Das A, Hale EC, Ball MB, Newman NS, Schibler K, Poindexter BB, Kennedy KA, Cotten CM, Watterberg KL, D'Angio CT, DeMauro SB, Truog WE, Devaskar U, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Trends in Care Practices, Morbidity, and Mortality of Extremely Preterm Neonates, 1993-2012. JAMA. 2015 Sep 8;314(10):1039-51. doi: 10.1001/jama.2015.10244. PMID 26348753
- [Background] Vardar-Yagli N, Inal-Ince D, Saglam M, Arikan H, Savci S, Calik-Kutukcu E, Ozcelik U. Pulmonary and extrapulmonary features in bronchopulmonary dysplasia: a comparison with healthy children. J Phys Ther Sci. 2015 Jun;27(6):1761-5. doi: 10.1589/jpts.27.1761. Epub 2015 Jun 30. PMID 26180315
- [Background] Vojta therapy in the reduction of perinatal risk in preterm infants with respiratory distress syndrome and bronchopulmonary dysplasia - Physiotherapy. (s. f.). Recuperado 1 de mayo de 2018, de https://www.physiotherapyjournal.com/article/S0031-9406(16)30315-7
- [Background] Zanudin A, Burns Y, Gray PH, Danks M, Poulsen L, Watter P. Perinatal events and motor performance of children born with ELBW and nondisabled. Pediatr Phys Ther. 2013 Spring;25(1):30-5. doi: 10.1097/PEP.0b013e31827aa424. PMID 23288005